CLINICAL TRIAL: NCT03004352
Title: Disturbed Blood Flow Induces Endothelial Dysfunction in Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Split, School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ED-COPD
Record Dates: First submitted 2016-12-20; First posted 2016-12-28 (Estimated); Last update posted 2016-12-28 (Estimated); Status verified 2016-12

CONDITIONS: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Oxygen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- control subjects-retrograde flow (Experimental): Retrograde flow was induced in control subjects.
  Interventions: Other: retrograde flow
- control subjects-control (No Intervention)
- hypoxemic COPD-retrograde flow (Experimental): Retrograde flow was induced in hypoxemic COPD patients.
  Interventions: Other: retrograde flow
- hypoxemic COPD-control (No Intervention)
- normoxemic COPD-retrograde flow with oxygen (Experimental): Retrograde flow was induced in COPD patients with normalized arterial oxygen saturation.
  Interventions: Other: retrograde flow; Other: oxygen
- normoxemic COPD-control with oxygen (Experimental): COPD patients with normalized arterial oxygen saturation.
  Interventions: Other: oxygen

INTERVENTIONS:
Other: retrograde flow — Two pneumatic cuffs were placed on the experimental arm, one on the lower forearm, and the other on the upper arm. Two cuffs were simultaneously inflated for 20 minutes. The distal cuff was inflated to 75 mm Hg and the proximal cuff was inflated to 40 mm Hg. The contralateral (control) arm was cuff free during this intervention.
  Arms: control subjects-retrograde flow; hypoxemic COPD-retrograde flow; normoxemic COPD-retrograde flow with oxygen
Other: oxygen — Supplemental 100% oxygen administered through a nasal cannula.
  Arms: normoxemic COPD-control with oxygen; normoxemic COPD-retrograde flow with oxygen

SUMMARY:
The aim of the study is to determine if increased retrograde shear would further deteriorate the already impaired vascular function in severe COPD patients.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* chronic hypoxemia

Exclusion Criteria:

* an acute exacerbation, active respiratory infection or infection of other localisation 6 weeks prior to the visit
* relevant coexisting lung disease such as interstitial lung disease, cancer, renal failure, thromboembolic disease or major cardiovascular event during the previous year
* informed consent not provided or inability to comply with the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-04; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Brachial Artery Diameter at 10, 20 and 25 minutes | 0,10, 20 and 25 minutes
Change from Baseline Microparticle Count at 20 minutes | 0 and 20 minutes

IPD SHARING:
Plan to Share IPD: No